CLINICAL TRIAL: NCT05792982
Title: Fluctuations of Serum Fibroblast Growth Factor-21 Levels During Prolonged Fasting in Male Adults
Brief Title: Serum Fibroblast Growth Factor-21 Levels During Prolonged Fasting
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Zeynep Goktas, Principal Investigator, Hacettepe University
Other Study IDs: GO 17/402
Record Dates: First submitted 2023-03-17; First posted 2023-03-31 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Fibroblast Growth Factor-21; Fasting
Keywords: FGF-21; Fasting; Ramadan
MeSH Terms: conditions — Fasting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples were collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fasting Adult Males: A questionnaire was administered in order to determine individuals' general characteristics, nutrition habits, and smoking and alcohol habits. Anthropometric measurements, 24 hours dietary recall and physical activities were recorded and blood samples were taken four times in following periods; before Ramadan, first week of Ramadan, third week of Ramadan and two weeks after Ramadan.
  Interventions: Behavioral: 12 hour fasting for 29 days

INTERVENTIONS:
Behavioral: 12 hour fasting for 29 days — This study aims to determine the effects of fasting on serum FGF21 levels. For this reason, male adults who fasted during the Ramadan were included in the study.

SUMMARY:
The investigators hypothesized that serum FGF21 levels would increase with prolongation of the fasting period. The investigators also hypothesized that food intake and body composition would change. The study was conducted with 12 healthy male adults. A questionnaire was administered at the beginning of the study. Anthropometric measurements, dietary intake and physical activities were recorded and blood samples were taken before, during and after Ramadan.

DETAILED DESCRIPTION:
The aim of this study was to determine the effects of hunger on serum Fibroblast Growth Factor 21 (FGF21) levels, nutritional status and anthropometric measurements of adult males during fasting. FGF21 is a significant protein in the process of adaption to fasting due to its effects on liver, adipose tissue, and brain. A total of 12 healthy individuals with normal body mass index, between the ages of 18 to 35 participated to this cross-sectional study. All participants provided written informed consent. Sample size determined with power analysis. A questionnaire was administered in order to determine individuals' general characteristics, nutrition habits, and smoking and alcohol habits. Anthropometric measurements, 24 hours dietary recall and physical activities were recorded and blood samples were taken four times in following periods; before Ramadan, first week of Ramadan, third week of Ramadan and two weeks after Ramadan. Serum FGF21 levels were determined by ELISA (Enzyme-Linked Immunosorbent Assay). Mean energy and nutrient intake were calculated by BEBIS (Nutrition Information System) and results were compared with Recommended Dietary Allowances (RDA). Paired samples t-test and Wilcoxon-signed rank test were used to explore differences. The study was approved by Hacettepe University Non-Interventional Clinical Research Ethics Board.

ELIGIBILITY:
Inclusion Criteria:

* Being healthy male,
* Being between the ages of 19-35,
* Fasting regularly during Ramadan.

Exclusion Criteria:

* Being females,
* Being younger than 19 years and older than 35 years of age,
* Having a BMI less than 18.5 kg/m2 and greater than 24.9 kg/m2,
* Having any chronic metabolic disease,
* Individuals who not fast regularly during Ramadan.

Ages: 19 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Individuals were recruited through social media announcements. Individuals residing in Ankara, where Hacettepe University is located, were recruited.
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-07-30 (Actual); Study Completion 2018-01-30 (Actual)

PRIMARY OUTCOMES:
FGF-21 levels | 3 months
  Blood samples were collected and serum FGF21 levels were determined by ELISA method
Body weight | 3 months
  Body weight was measured using a scale with 100g sensitivity.
Body fat ratio | 3 months
  Body fat ratio was measured by a bioelectrical impedance analysis device.
Body muscle composition | 3 months
  Body fat composition was measured by a bioelectrical impedance analysis device.
Dietary Intake | 3 months
  24-hour dietary recall questionnaires were administered by researchers.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Goktas, PhD, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University Nutrition and Dietetics Department, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No